CLINICAL TRIAL: NCT04863105
Title: Bioequivalence of Abiraterone Acetate in Healthy Chinese Volunteers: an Open, Randomized, Single-dose, Three-cycle, Three-sequence Crossover Study
Brief Title: Bioequivalence of Abiraterone Acetate Tablets in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: QL-YK4-047-001
Record Dates: First submitted 2021-03-23; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: an open, randomized, single-dose, three-cycle, three-sequence crossover study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conference-Abiraterone acetate tablet (Experimental): Abiraterone acetate tablets(Zecke ® 250 mg,Batch number:VYCB manufactured by Patheon Inc.)
  Interventions: Drug: Abiraterone acetate tablets(Zecke ®250 mg);Abiraterone acetate tablets(250 mg)
- test-Abiraterone acetate tablet (Experimental): Abiraterone acetate tablets(250 mg,Batch number:17F0023DD9 manufactured by Qilu Pharmaceutical Co., Ltd)
  Interventions: Drug: Abiraterone acetate tablets(Zecke ®250 mg);Abiraterone acetate tablets(250 mg)

INTERVENTIONS:
Drug: Abiraterone acetate tablets(Zecke ®250 mg);Abiraterone acetate tablets(250 mg) — Subjects were allocated to one of three groups randomly and equally with a 7-day washout interval between the two periods."Abiraterone acetate tablets(Zecke ® 250 mg,Batch number:VYCB manufactured by Patheon Inc.)and Abiraterone acetate tablets(250 mg,Batch number:17F0023DD9 manufactured by Qilu Pharmaceutical Co., Ltd) were used in this study.

SUMMARY:
An open, randomized, single-dose, three-cycle, three-sequence crossover study was conducted in 36 healthy volunteers under fasting condition to evaluate the bioequivalence of two abiratone acetate tablets.

DETAILED DESCRIPTION:
Abiraterone acetate tablet is an androgen synthesis inhibitor, primarily for the treatment of mCRPC. The objective of this study was to evaluate the pharmacokinetics and bioequivalence of two abiraterone acetate tablets in healthy Chinese subjects. In healthy subjects, a single-center, open, single-dose, randomized, three-cycle, three-sequence, semi-repeat (duplicate reference preparation only), reference formulation corrected fasting mean bioequivalence trial was conducted with a minimum of 7 days cleaning period between dosing.

Blood samples were collected at prescribed time intervals, and the plasma concentration of abiraterone acetate tablet was determined by liquid chromatography-tandem mass spectrometry and adverse events were recorded.

The pharmacokinetic parameters Cmax, Tmax, AUC0-t, AUC0-∞, T1/2 and so on were calculated by non-atrioventricular model. When the individual coefficient of variation(CVWR) of the pharmacokinetic parameters (AUC0-t, AUC0-∞ and Cmax) of reference formulation was less than 30%,with an average bioequivalence (ABE) criterion: if the test formulation and reference formulation of pharmacokinetic parameters (AUC0 - t,AUC0-∞ and Cmax) of the 90% CIs of GMR is not beyond the range of 80.00% -125.00%, which can determine the test formulation and reference formulation have bioequivalence.When the CVWR of the pharmacokinetic parameters (AUC0-t, AUC0-∞ and Cmax) of the reference preparation is greater than or equal to 30%,the reference preparation was used to correct for mean bioequivalence (RSABE): if the critbound of the pharmacokinetic parameters (AUC0-t,AUC0-∞ , Cmax) of the test formulations and reference formulations is less than 0, and the geometric average ratio is not beyond the range of 0.8000 - 1.2500, which can determine the test formulation and reference formulation have bioequivalence.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects above 18 years old (including 18 years old).
* Weight not less than 50 kg, body mass index between 19 and 28kg/m2.
* No bad habits such as smoking or alcohol, and no history of drug abuse.
* Subjects are willing to have no birth plan in the next 6 months and voluntarily take effective contraceptive measures.
* Volunteered to participate in the clinical trial, understood the study procedures and signed the written informed consent. Able to complete the study according to the test protocol.

Exclusion Criteria:

* Abnormal results of vital signs, physical examination, electrocardiogram and other laboratory examinations were clinically significant.
* With the central nervous system, cardiovascular system, liver and kidney function is not complete, the digestive system (not included in the drug delivery two weeks ago suffering from acute gastroenteritis, diarrhea), respiratory system (not included in the drug delivery two weeks ago with upper respiratory infection), metabolism and skeletal system disease, or any other may affect the results of the study of disease and physiological conditions.
* A history of hospitalization or surgery within 3 months prior to the trial.
* Known active hepatitis B, HIV, HCV and Treponema pallidum infection.
* Have a history of specific allergic reactions (such as atopic dermatitis, asthma, etc.), or have a history of allergy to drugs and biological agents, or have a history of known allergy to the ingredients of this drug.
* Positive alcohol and urine drug screening.
* Regular drinkers who consumed more than 14 units of alcohol per week (1 unit is 360 mL beer or 45 mL liquor of 40% alcohol or 150 mL wine) during the 3 months prior to the trial.
* Smoking more than 5 cigarettes per day within 3 months before the trial.
* Participate as a subject in any drug clinical trial within 3 months prior to the trial.
* People who had donated blood or lost more than 400mL of blood in 3 months before the experiment.
* Have taken any prescription drugs during the 14 days prior to the trial. Have taken any over-the-counter medicines, any functional vitamins or herbal products within 48 hours prior to the trial.
* Have consumed any xanthine-rich beverage or food or grapefruit fruit or products containing grapefruit within 48 hours prior to the test.
* Have consumed any food or drink containing caffeine (such as tea or coffee) and any alcoholic products within 48 hours before the trial.
* Have special requirements on diet and fail to follow the diet and corresponding regulations provided.
* Subjects who are considered by the investigator to have poor compliance or have any unsuitable factors for participating in the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2017-12-25 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
the ratios of geometrical mean | 30 Days
  The two formulations are considered to be bioequivalent if the CVWR is less than 30% and 90% CIS of the ratio of primary pharmacokinetic parameters is within a predetermined acceptance range of 80% to 125%. If the CVWR of the pharmacokinetic parameters of the reference preparation is greater than or equal to 30%, Critbound ≤0, and the geometric mean ratio does not exceed the range of 0.8000 to 1.2500, the test preparation and the reference preparation can be determined to be bioequivalent.

SECONDARY OUTCOMES:
the occurrence rate of adverse events | 30 Days
  Adverse events were recorded to evaluate the safety of the studied drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, Doctor, Principal Investigator — the study director of phase I clinical research center
Locations (1):
- Phase I Clinical Research Center, Qingdao, Shangdong, China

IPD SHARING:
Plan to Share IPD: No
All the technical achievements and outcomes of this trial are owned by Qilu Pharmaceutical Co., Ltd. and the research center. The research center can not publish any academic papers without the consent of the sponsor.

REFERENCES:
- [Derived] Wu ZX, Wang CJ, Shi P, Liu YP, Li T, Sun FF, Fu Y, Gao XM, Ma YP, Cao Y. Pharmacokinetics and Bioequivalence of Abiraterone Acetate Tablets in Healthy Chinese Volunteers: An Open, Randomized, Single-Dose, Three-Period, Three-Sequence Crossover Study. Drugs R D. 2023 Jun;23(2):121-127. doi: 10.1007/s40268-023-00418-6. Epub 2023 Apr 3. PMID 37012461